CLINICAL TRIAL: NCT05430477
Title: Characterizing In Vivo Oral Lesion Impedances
Status: Completed | Type: Observational
Sponsor: Ryan J. Halter (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Dartmouth College (Other)
Responsible Party: Sponsor-Investigator, Ryan J. Halter, Investigator and Regulatory Sponsor, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Other Study IDs: STUDY02001317; R21DE031095-01 (NIH)
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Oral Lesion
Keywords: electrical impedance tomography (EIT); Oral Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1 Biopsy: Subjects recruited to Cohort I will include patients who are scheduled to undergo oral lesion biopsy as well as patients who are determined to need a biopsy at the time of visual examination, which often occurs in-clinic. Cohort I will consist of 125 oral lesion biopsy patients total. Prior to the start of enrollment in this Cohort, up to 5 additional subjects will be enrolled to optimize the data acquisition process.
  Interventions: Device: Electrical impedance imaging using Non-Significant Risk device (EII probe)
- Cohort 2 Resection: Potential study participants will be identified through Dartmouth-Hitchcock Medical Center (DHMC)'s Head and Neck Tumor Clinic, and will be patients with diagnosed or suspected cancer of the oral cavity, oropharynx, hypopharynx, or larynx who require biopsy or resection for either diagnostic or therapeutic purposes. Cohort II will be comprised of 125 patients undergoing oral cavity cancer resections. Initially, up to 5 subjects will be enrolled in addition to the 125 patients in this Cohort in order to optimize the data acquisition process.
  Interventions: Device: Electrical impedance imaging using Non-Significant Risk device (EII probe)

INTERVENTIONS:
Device: Electrical impedance imaging using Non-Significant Risk device (EII probe) — novel small field-of-view Non-Significant Risk device (EII probe)

SUMMARY:
The primary objective of this study is to demonstrate a significant difference in electrical impedance between normal, benign, premalignant, and malignant oral lesions using a custom device. The secondary study objective is to create a database of in vivo electrical impedance spectra and images of oral lesions. This will be achieved by collecting Electrical Impedance sensing data and images from two cohorts of patients: Cohort I will consist of 200 patients undergoing oral lesion biopsies and Cohort II will be comprised of 50 patients scheduled for oral cancer resection. A maximum of 5 additional subjects will be initially enrolled in each Cohort to optimize data acquisition.

DETAILED DESCRIPTION:
For this study, a novel small field-of-view EII probe will be used for recording impedances from oral lesions. The device is comprised of gold-plated electrodes with analog electronics located in the probe's tip, to minimize cable lengths and maximize the signal-to-noise ratio. A pressure sensor is embedded within the probe to reduce variability in the amount of pressure used when the probe is applied to soft tissue. The bioimpedance-sensing probe is designed to the following specifications in order to accurately assess oral lesions:

1. measurement precision ~85 dB,
2. accuracy >99%,
3. bandwidth extending to 1 MHz, and
4. multi-frequency sample rate of >10 impedance spectra per second.

Similar to other EII systems the team has developed and deployed in vivo, the system complies with International Electrotechnical Commission (IEC) requirements for safety and essential performance of medical electrical equipment (IEC 60601-1).

There are no known probes cleared by the FDA for this application.

The study is not being conducted in order to evaluate the EII probe's safety or effectiveness in human subjects, nor to test the device for marketing or promotion.

ELIGIBILITY:
Cohort 1 10.1.1 Inclusion Criteria

1. Suspected cancer the oral cavity, oropharynx, hypopharynx, or larynx requiring biopsy.
2. Ability to understand and the willingness to sign a written informed consent document.
3. Age ≥ 18 years old.
4. If a female of child bearing potential, then a negative pregnancy evaluation per standard of care.

10.1.2 Exclusion Criteria

1. Adults having had a previous oral biopsy within the last 30 days
2. Adults with implanted electrical devices such as pacemakers
3. Prisoners
4. Adults with impaired decision-making capacity
5. Has any condition for which, in the opinion of the investigator, contraindicates study participation.

Cohort 2 10.2.2 Inclusion Criteria

1. Clinical diagnosis or suspected cancer the oral cavity, oropharynx, hypopharynx, or larynx requiring resection.
2. Ability to understand and the willingness to sign a written informed consent document.
3. Age ≥ 18 years old
4. If a female of child bearing potential, then a negative pregnancy evaluation per standard of care.

10.2.3 Exclusion Criteria

1. Adults with implanted electrical devices such as pacemakers
2. Prisoners
3. Adults with impaired decision-making capacity
4. Any condition for which, in the opinion of the investigator, contraindicates study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be identified through Dartmouth-Hitchcock Medical Center (DHMC)'s Head and Neck Tumor Clinic, and will be patients with diagnosed or suspected cancer of the oral cavity, oropharynx, hypopharynx, or larynx who require biopsy or resection for either diagnostic or therapeutic purposes. This study will enroll 250 subjects in two cohorts. Cohort I will consist of 200 patients undergoing oral lesion biopsies. Cohort II will be comprised of 50 patients scheduled for oral cancer resection. A maximum of 5 additional subjects will be initially enrolled in each Cohort to optimize data acquisition.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Differences in Electrical Impedance | Participants are on study only the day of the procedure.
  This study will use a custom device to measure differences in electrical impedance between normal, benign, premalignant, and malignant oral lesions.

SECONDARY OUTCOMES:
Images and Measurements Database Creation | Participants are on study only the day of the procedure.
  Images and in vivo electrical impedance spectra measurements taken for each participant on the day of the procedure will be used to create a database.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Halter, PhD, Principal Investigator — Trustees of Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States